CLINICAL TRIAL: NCT06803290
Title: An Open-Label, Two-Period, Two-Sequence, Two-Treatment Randomized, Single Oral Dose, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetic Profile of VHX-896 in Healthy Volunteers
Brief Title: Food Effect Study of VHX-896 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VP-VHX-896-1102
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: VHX-896; Food Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: fed then fasted (Experimental)
  Interventions: Drug: VHX-896
- Sequence B: fasted then fed (Experimental)
  Interventions: Drug: VHX-896

INTERVENTIONS:
Drug: VHX-896 — Oral tablet

SUMMARY:
A single center, two-period, randomized study to evaluate the food effect of VHX-896 tablets in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants between 18 to 55 years (inclusive).
* Have a Body Mass Index (BMI) of > 18.0 and < 30.0 kg/m2; (BMI = weight (kg)/ [height (m)]2).
* Good health as determined by no clinically significant deviations from normal in medical history, clinical laboratory determination, ECGs, and physical examinations.
* No clinically significant medical, psychiatric or sleep disorders.

Exclusion Criteria:

* Participants with history of drug or alcohol abuse in last 12 months.
* Participants who suffered from significant physical illness in the 4-week period preceding baseline.
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Comparative bioavailability of VHX-tablets under fed versus fasted conditions. | 96 Hours
  As measured by plasma concentrations

SECONDARY OUTCOMES:
Assessment of safety and tolerability of single dose of VHX-896 tablets | 17 Days
  As measured by the incidence of adverse events and clinically significant changes in laboratory values, ECG parameters, and vital signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No